CLINICAL TRIAL: NCT06685016
Title: Evaluation of Dental and Periodontal Health After Interproximal Enamel Reduction, in Patients in Orthodontic Treatment With Clear Aligners, and Comparison Between Laser Diode and Sodium Fluoride for the Treatment of Dentin Hypersensitivity
Brief Title: Evaluation of Dental and Periodontal Health After IPR in Patients in Orthodontic Treatment With Clear Aligners
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Vincenzo Grassia, Associate Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 0016945/i
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Dentinal Hypersensitivity; Plaque, Dental; Bleeding Gum
Keywords: Clear Aligners; Interproximal enamel reduction
MeSH Terms: conditions — Dental Plaque; Gingival Hemorrhage

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Experimental): Subjects will not receive any treatment
  Interventions: Diagnostic Test: Evaluation of Dentin hypersensitivity with VAS scale
- Laser Diode Group (Experimental): Subjects treated with Laser Diode
  Interventions: Diagnostic Test: Evaluation of Dentin hypersensitivity with VAS scale
- Sodium Fluoride Group (Experimental): Subjects with a sodium fluoride gel treatment.
  Interventions: Diagnostic Test: Evaluation of Dentin hypersensitivity with VAS scale

INTERVENTIONS:
Diagnostic Test: Evaluation of Dentin hypersensitivity with VAS scale — Dentin hypersensitivity and periodontal indices evaluation are performed after and before IPR, at 1 week, 1 month and 3 months

SUMMARY:
This study aimed to evaluate dental and periodontal health after interproximal enamel reduction and to compare Laser diode (a device used in the Orthodontic Program) and sodium fluoride (often used in the Orthodontic Program and in the Material Dental Program). The hypothesis was that the intervention groups would show a lower dentin hypersensitivity incidence than the control group during orthodontic treatment.

DETAILED DESCRIPTION:
Interproximal enamel reduction (IPR) is a common procedure used during orthodontic treatment aimed to reduce mesio-distal tooth size dimensions to address lack of space (mild and moderate crowding), Bolton tooth-size discrepancy, correction of morphologic anomalies, tooth reshaping and management of gingival papilla. It is a practice that also offers an attractive alternative to overcome difficulty when extracting premolars and resolve the instability of overexpansion in non- extraction cases, improving the stability of the arches.

IPR may be exploited inconjunction with fixed appliance treatment, although its application with removable appliance treatment such as clear aligners is commonplace.

Clinically, the most accepted IPR techniques include air-rotor stripping with fine tungsten-carbide or diamond burs, handpiece or contra-angle-mounted diamond-coated disks, and handheld or motor- driven abrasive metal strips.

Some of these techniques can cause deep furrows and scratches that cannot be removed by polishing . In addition, these surface irregularities could promote the adherence of plaque bacteria and induce iatrogenic damage, such as dental caries, gingival inflammation, periodontal tissue breakdown, gingival recession and increased sensitivity of the shaped teeth to hot and cold temperatures.

Sometimes, after IPR, it is possible to have dentin hypersensitivity (DH), attributed to exposure to dentinal tubules. This clinical condition is influenced by various factors, including patient' s age, the severity of crowding, pathological tooth wear, hypersensitivity before treatment and the amount of the removed enamel.

DH can be defined as "short and sharp pain due to exposure of the dentinal tubules in response to thermal, evaporative, tactile, osmotic or chemical stimuli". The hydrodynamic theory proposed by Brännström is the most accepted theory to explain the DH mechanism. According to this theory, external stimuli, leading to fluid movement within the dentinal tubules and this movement indirectly stimulates the pulp nerve ends, causing a painful sensation.

Several methods can perform DH treatment. Based on the mode of their administration, the desensitizing treatment can be classified into at-home therapy or in-office therapy categories. At- home desensitizing products include toothpaste, mouthwashes and chewing gums. In contrast, in- office desensitizing products can be gels, solutions, varnishes, resin sealers, glass ionomers, dentin adhesives and more sophisticated laser techniques. In addition, eliminating of nociceptive stimuli, there are two main treatment strategies: modifying nervous response by preventing or reducing neuronal transmission and occluding the permeable dentinal tubules.

Potassium salts were thought to decrease the excitability of pulpal nerves and result in a reduction in DH. Still, clinical trials with sound design have failed to provide evidence that potassium is effective in desensitizing teeth. Potassium salts likely reduced the perception of dentin sensitivity through a placebo effect. The proposed mechanism for glutaraldehyde, another agent used for the treatment of DH, involves the reaction with serum albumin in dentinal tubule fluid, leading to precipitate formation within tubules and subsequent narrowing or blocking of the tubules. Strontium salts, fluoride, oxalate and arginine/calcium can occlude the tubules and form a protective layer on the dentin surface. Dental adhesives and resin sealants can occlude the dentinal tubules by forming a physical barrier thus blocking the movement of dentinal fluid and preventing direct stimulation of odontoblastic processes. The action of glass ionomers in the management of DH can also lead to occlusion of open dentinal tubules by precipitating a hydroxycarbonate apatite layer over the previously patent tubule openings. Laser treatment has been investigated as a prospective treatment for DH. Several studies suggest that the low-power laser could suppress the excitability of the pulpal nerves. Higher output laser is thought to reduce symptoms of DH by inducing the occlusion of dentin tubules.

Pain associated with DH may reduce the quality of life, but does not compromise people's health. Currently, no studies that have tested desensitizing substances to reduce or eliminate DH that can occur after IPR.

ELIGIBILITY:
Inclusion Criteria:

* to be in orthodontic treatment with clear aligners and this treatment requires interproximal enamel reduction;
* permanent dentition;
* good oral and periodontal health.

Exclusion Criteria:

* enamel defects;
* cervical caries;
* periodontal disease;
* history of trauma or craniofacial anomalies;
* pregnancy.

Ages: 17 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Assestment of DH after IPR | from 3 to 4 months
  Dentin hypersensitivity will be assessed before and after interproximal enamel reduction and after the application of therapeutic protocols. Dentin hypersensitivity will be performed with the evaporative method. After isolation of the adjacent teeth, the air syringe will be placed 2-3 mm from the tooth surface, at a perpendicular position of 90º, and a continuous air blast of 45 to 60 psi (3.10 to 4.13 Bar) should be applied for 2-3 seconds. The air temperature should be around 20°C (19-22°C). The discomfort will be expressed in a numerical 0-10 cm visual analog scale (VAS) where the value 0 is correlated with no discomfort and the value 10 for utmost discomfort or intolerable pain during application of the stimulus. Each patient will place a vertical mark on the VAS to indicate the intensity of his or her level of sensitivity after the applied stimuli.
Reduction of the Dentin Hypersensitivity | from 3 to 4 months
  . Dentin hypersensitivity will be performed with the evaporative method. After isolation of the adjacent teeth, the air syringe will be placed 2-3 mm from the tooth surface, at a perpendicular position of 90º, and a continuous air blast of 45 to 60 psi (3.10 to 4.13 Bar) should be applied for 2-3 seconds. The air temperature should be around 20°C (19-22°C). The discomfort will be expressed in a numerical 0-10 cm visual analog scale (VAS) where the value 0 is correlated with no discomfort and the value 10 for utmost discomfort or intolerable pain during application of the stimulus. Each patient will place a vertical mark on the VAS to indicate the intensity of his or her level of sensitivity after the applied stimuli.

SECONDARY OUTCOMES:
Evaluation of Dentin hypersensitivity after the application of therapeutic protocols. | from 3 to 4 months
  Evaluate Dentin Hypersensitivity in the control group and the treated groups,with the evaporative method. After isolation of the adjacent teeth, the air syringe will be placed 2-3 mm from the tooth surface, at a perpendicular position of 90º, and a continuous air blast of 45 to 60 psi (3.10 to 4.13 Bar) should be applied for 2-3 seconds. The air temperature should be around 20°C (19-22°C). The discomfort will be expressed in a numerical 0-10 cm visual analog scale (VAS) where the value 0 is correlated with no discomfort and the value 10 for utmost discomfort or intolerable pain during application of the stimulus. Each patient will place a vertical mark on the VAS to indicate the intensity of his or her level of sensitivity after the applied stimuli.
  To assess in which group it reduces or is eliminated more quickly.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Grassia, DDs,PhD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Multidisciplinary department of Medical-Surgical and Dental Specialties, Naples, Italy

REFERENCES:
- [Background] Liu XX, Tenenbaum HC, Wilder RS, Quock R, Hewlett ER, Ren YF. Pathogenesis, diagnosis and management of dentin hypersensitivity: an evidence-based overview for dental practitioners. BMC Oral Health. 2020 Aug 6;20(1):220. doi: 10.1186/s12903-020-01199-z. PMID 32762733
- [Background] Poulsen S, Errboe M, Lescay Mevil Y, Glenny AM. Potassium containing toothpastes for dentine hypersensitivity. Cochrane Database Syst Rev. 2006 Jul 19;2006(3):CD001476. doi: 10.1002/14651858.CD001476.pub2. PMID 16855970
- [Background] Orchardson R, Gillam DG. The efficacy of potassium salts as agents for treating dentin hypersensitivity. J Orofac Pain. 2000 Winter;14(1):9-19. PMID 11203743
- [Background] Livas C, Jongsma AC, Ren Y. Enamel reduction techniques in orthodontics: a literature review. Open Dent J. 2013 Oct 31;7:146-51. doi: 10.2174/1874210601307010146. eCollection 2013. PMID 24265652
- [Background] Boyd RL. Esthetic orthodontic treatment using the invisalign appliance for moderate to complex malocclusions. J Dent Educ. 2008 Aug;72(8):948-67. PMID 18676803
- [Background] Pindoria J, Fleming PS, Sharma PK. Inter-proximal enamel reduction in contemporary orthodontics. Br Dent J. 2016 Dec 16;221(12):757-763. doi: 10.1038/sj.bdj.2016.945. PMID 27982013
- [Background] Lombardo L, Guarneri MP, D'Amico P, Molinari C, Meddis V, Carlucci A, Siciliani G. Orthofile(R): a new approach for mechanical interproximal reduction : a scanning electron microscopic enamel evaluation. J Orofac Orthop. 2014 May;75(3):203-12. doi: 10.1007/s00056-014-0213-0. Epub 2014 May 15. PMID 24825832
- [Background] Joseph VP, Rossouw PE, Basson NJ. Orthodontic microabrasive reproximation. Am J Orthod Dentofacial Orthop. 1992 Oct;102(4):351-9. doi: 10.1016/0889-5406(92)70051-B. PMID 1333728
- [Background] Zachrisson BU. Actual damage to teeth and periodontal tissues with mesiodistal enamel reduction ("stripping"). World J Orthod. 2004 Summer;5(2):178-83. No abstract available. PMID 15615137
- [Background] Jarjoura K, Gagnon G, Nieberg L. Caries risk after interproximal enamel reduction. Am J Orthod Dentofacial Orthop. 2006 Jul;130(1):26-30. doi: 10.1016/j.ajodo.2004.08.024. PMID 16849068
- [Background] Lapenaite E, Lopatiene K. Interproximal enamel reduction as a part of orthodontic treatment. Stomatologija. 2014;16(1):19-24. PMID 24824056
- [Background] Marto CM, Baptista Paula A, Nunes T, Pimenta M, Abrantes AM, Pires AS, Laranjo M, Coelho A, Donato H, Botelho MF, Marques Ferreira M, Carrilho E. Evaluation of the efficacy of dentin hypersensitivity treatments-A systematic review and follow-up analysis. J Oral Rehabil. 2019 Oct;46(10):952-990. doi: 10.1111/joor.12842. Epub 2019 Jul 12. PMID 31216069